CLINICAL TRIAL: NCT03009045
Title: Tolerability, Safety, and Efficacy of Tedizolid as Oral Treatment for Bone and Joint Infections
Brief Title: Tolerability, Safety, and Efficacy of Tedizolid as Oral Treatment for Bone and Joint Infections (OTTER)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, loren g miller, Primary Investigator, Associate Chief of Division of Infectious Diseases, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21814-01
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Bone and Joint Infection
Keywords: bone and joint infection; osteomyelitis; tedizolid
MeSH Terms: conditions — Osteomyelitis | interventions — tedizolid; tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: 200mg oral Tedizolid (Experimental): 200mg oral tablet of tedizolid to be taken once daily
  Interventions: Drug: Tedizolid

INTERVENTIONS:
Drug: Tedizolid — 200mg oral tedizolid one pill per day
  Other Names: tedizolid phosphate; Sivextro

SUMMARY:
The problem of interest is that doctors are looking for new antibiotic treatments for bone and joint infections. Treatment for bone and joint infection is not standardized, which allows a wide range of antibiotic therapy to potentially be given. A type of bacteria called S. aureus is the most common cause of bone and joint infection. Methicillin resistant S. aureus (MRSA) is a type of bacteria that is not killed by some antibiotics, and it is increasingly common in U.S. and non-U.S. medical centers. This problem will be studied by investigating whether an antibiotic called tedizolid is tolerable, safe and effective to treat bone and joint infections.

DETAILED DESCRIPTION:
The problem of interest is that doctors are looking for new antibiotic treatments for bone and joint infections. Treatment for bone and joint infection is not standardized, which allows a wide range of antibiotic therapy to potentially be given. A type of bacteria called S. aureus is the most common cause of bone and joint infection. Methicillin resistant S. aureus (MRSA) is a type of bacteria that is not killed by some antibiotics, and it is increasingly common in U.S. and non-U.S. medical centers. Trauma-associated bone and joint infection is also a common problem. Victims of major trauma often suffer bone fractures, which require temporary or permanent use of metal or other synthetic devices such as external-fixation pins, plates, and screws. These synthetic devices can also get infected and cause bone and joint infections.

This problem will be studied by investigating whether an antibiotic called tedizolid is tolerable, safe and effective to treat bone and joint infections. Tedizolid is a new FDA-approved antibiotic, and can be given through the bloodstream via an IV or orally in the form of a pill. Tedizolid has less side effects compared to linezolid and is effective against types of bacteria like S. aureus. Other research also suggests that the side effects associated with long-term therapy of older types of antibiotics may not be found with tedizolid.

This study will advance scientific knowledge of antibiotic treatments for bone and joint infections. Given the large and increasing burden of disease of bone and joint infection and the increasing acceptability of oral antibiotics for its management, tedizolid holds promise as a good option for patients with bone and joint infection. Harbor-UCLA Medical Center is a large medical center in the County of Los Angeles, the most populous County in the United States. The Infectious Disease consult service sees many bone and joint infections. Use of prolonged antibiotics is common in this setting. The investigators believe tedizolid addresses the unmet need for an oral antibiotic that is well-tolerated and efficacious for use as a prolonged therapy for bone and joint infection.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of bone and joint infection in which therapy for Gram positive organisms is documented or suspected, as determined by the treating physician and treatment of at least 4 weeks is planned. Bone and joint infection and trauma-associated bone and joint infection will defined clinically using radiologic (e.g., MRI) and/or surgical (e.g., intra-operative findings) definitions. All subjects must have confirmation (diagnosis mentioned in chart) by the patient's primary physician and consultants that the patients has or likely has bone and joint infection and requires prolonged antibiotic therapy.
* Aged between 18 years and 85 years.
* Plans to treat bone and joint infection in outpatient setting.
* No limited planned course of antibiotics (i.e., no indefinite treatment plans for chronic suppression). Co-administration of other antibiotics that target other causative or potentially causative organisms (e.g., fluoroquinolones) is acceptable.
* Able to come to the research clinic for study follow-up visits for the study period.

Exclusion Criteria:

* Planned prolonged hospitalization (> 1 week).
* Pregnancy (all female subjects of childbearing age will be given a pregnancy test prior to enrollment) or breast feeding. If a women is of childbearing potential, she must consistently use an acceptable method of contraception (IUD, injectable contraceptive, birth control patch, OCP, barrier method, abstinence) from baseline through the course of antibiotics (4-12 weeks). If a male patient's sexual partner is of childbearing potential, the male patient must acknowledge that they will consistently use an acceptable method of contraception as defined above from baseline through the course of antibiotics (4-12 weeks).
* Comorbidities that, in the opinion of the investigator, are uncontrolled (e.g., diabetes, hypertension, psychiatric disease).
* Peripheral or optic neuropathy.
* Underlying hematologic cytopenias (e.g., baseline thrombocytopenia, or severe anemia, or leukopenia) as determined by the following limits from a baseline CBC/CMP obtained within the past 14 days. Note that if a CBC has not been performed within the past 14 days, a CBC will be performed on the day of enrollment prior to any study drug being administered to ensure the patient does not meet exclusion criteria. Cytopenias are defined as:

  1. Hemoglobin (Hgb) < 8.0g/dL
  2. WBC < 4,000 k/cumm
  3. Platelets < 150,000 k/cumm
* Severe hepatic dysfunction as defined by liver function tests (ALT, ALP, AST, total bilirubin) > 3.0 times the upper limit of normal. as determined by the following limits from a baseline CMP obtained within the past 7 days. If a CMP has not been performed within the past 7 days, baseline levels may be used from a CMP performed within the past 2 months as long as another CMP is performed on the day of enrollment and the subject's levels are within the following limits.
* Hypersensitivity to tedizolid or other oxazolidinone-class antibiotics or similar compounds.
* Ongoing antibiotic-associated colitis.
* A diet high in tyramine-containing foods such as pickled or fermented meats and cheeses, wine, or avocados per investigator discretion.
* Concurrent use of sodium picosulfate (brand names: Sodipic Picofast, Laxoberal, Laxoberon, Purg-Odan, Picolax, Guttalax, Namilax, Pico-Salax and Prepopik).
* Previous participation in the study.
* Use of tedizolid for any condition in the past 3 months.
* Any other medical, psychological, or social condition that, in the opinion of the Investigator, would prevent the patient from fully participating in the study or would represent a concern for study compliance or constitute a safety concern to the patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren G Miller, MD MPH, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (2):
- United States (2):
  - Harbor-UCLA Medical Center, Torrance, California
  - Los Angeles BioMedical Research Institute (LA BioMed), Torrance, California

IPD SHARING:
Plan to Share IPD: Yes
After publication of trial results, data will be shared with investigators upon request to the Principal Investigator and after signing a Data Use Agreement.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Miller LG, Flores EA, Launer B, Lee P, Kalkat P, Derrah K, Agrawal S, Schwartz M, Steele G, Kim T, Kuvhenguhwa MS. Safety and tolerability of tedizolid as oral treatment for bone and joint infections. Microbiol Spectr. 2023 Sep 26;11(5):e0128223. doi: 10.1128/spectrum.01282-23. Online ahead of print. PMID 37750695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: 200mg Oral Tedizolid
Started | 44
Completed | 37
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Not different from assignment in participant flow
Arm/Group | Drug: 200mg Oral Tedizolid
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 46 [22 to 65]
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean | 44 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 23
  White | 2
  Black/African American | 10
  Native American/Native Indian | 1
  Decline to State | 1
Region of Enrollment [Number; unit: participants]
  United States | 37
Type of Bone or Joint Infection [Number; unit: participants]
  Hardware-associated infection | 17
  Osteomyelitis, non-hardware associated | 13
  Prosthetic joint infection | 5
  External-fixator associated | 1
  Septic arthritis | 1

OUTCOME MEASURES:

1. Primary Outcome: Quantify the Tolerability of Tedizolid for Bone and Joint Infections, Both Hardware and Non-hardware Associated
Description: Tolerability was measured by interview. We asked participants weekly about new symptoms that could suggest new onset of peripheral or optic neuropathy.
Time Frame: 4-12 Weeks
Measure: Number; unit: participants
Arm/Group | Drug: 200mg Oral Tedizolid
Number analyzed (Participants) | 37
participants
  Reported peripheral neuropathy | 0
  Reported optic neuropathy | 0

2. Primary Outcome: Quantify the Safety of Tedizolid for Bone and Joint Infections, Both Hardware and Non-hardware Associated
Description: Safety, was measured by weekly complete blood counts (CBC), and comprehensive metabolic panels (CMP) were performed.
Time Frame: 4-12 Weeks
Measure: Number; unit: participants
Arm/Group | Drug: 200mg Oral Tedizolid
Number analyzed (Participants) | 37
participants
  High leukocytes | 0
  Low leukocytes | 0
  Low hemoglobin | 0
  Low plateltes | 0
  High AST | 0
  High ALT | 0
  High ALP | 0

3. Other Pre Specified Outcome: Number of Participants With an Outcome of "Cure" as Defined as no Need for Further Antibiotics Beyond the Originally Planned Duration Determined by the Participant's Primary/Treating Physician.
Description: Study Hypothesis: Tedizolid is effective for the treatment of bone and joint infection. Specifically, cure will be defined as no need for further antibiotics beyond the originally planned duration (i.e., 6 weeks for non-device associated bone and joint infection or until hardware removal for subjects with implants). Unplanned surgical procedures prompted by inadequate infection control will be categorized as treatment failure. We will also measure long-term cure by performing a phone survey 3 months after completion of antibiotics. Recurrence of signs or symptoms of bone and joint infection will be considered not a long-term treatment cure (i.e., failure).
Time Frame: 16-24 Weeks
Measure: Number; unit: participants
Arm/Group | Drug: 200mg Oral Tedizolid
Number analyzed (Participants) | 37
participants | 13

ADVERSE EVENTS:
Time Frame: 16 weeks to 24 weeks
Arm/Group | Drug: 200mg Oral Tedizolid
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 2/44
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: 200mg Oral Tedizolid (N=44)
Rash (Skin and subcutaneous tissue disorders) | 2 — Self-limited non-life threatening maculopapular rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03009045/Prot_SAP_000.pdf